CLINICAL TRIAL: NCT01782898
Title: The Effect of Intraoperative Esmolol to Improve Postoperative Quality of Recovery and Pain After Ambulatory Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Prinipal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00066623
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: Anesthesia; MEDOC neuro sensory analyzer; Pain; Quality of recovery
MeSH Terms: conditions — Pain | interventions — esmolol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esmolol (Active Comparator): Esmolol administered at a rate of 0.5 mg/kg followed by an infusion of 5-15 mcg/kg/min
  Interventions: Drug: Esmolol administered at a rate of 0.5 mg/kg followed by an infusion of 5-15 mcg/kg/min
- .9 normal saline (Placebo Comparator): .9 normal saline infused at the same rate (/mg/kg bolus followed by 5-15 mcg/kg/mn) as the Esmolol would be administered,
  Interventions: Drug: Placebo Comparator: .9 normal saline

INTERVENTIONS:
Drug: Esmolol administered at a rate of 0.5 mg/kg followed by an infusion of 5-15 mcg/kg/min — Esmolol administered at a rate of 0.5 mg/kg followed by an infusion of 5-15 mcg/kg/min
  Other Names: Esmolol
  Arms: Esmolol
Drug: Placebo Comparator: .9 normal saline — Placebo Comparator: Placebo .9 normal saline infused at the same rate (/mg/kg bolus followed by 5-15 mcg/kg/mn) as the Esmolol would be administered,
  Other Names: Normal Saline
  Arms: .9 normal saline

SUMMARY:
Seventy percent of surgeries performed in the United States are done in an outpatient setting.Pain Control after ambulatory surgery is very challenging because patients do not have access to fast and potent intravenous medications Pain after ambulatory surgery is poorly controlled in the United States with up to seventy five percent of patients having moderate to severe pain after ambulatory procedures. Postoperative pain have been associated with serious morbidity, including myocardial infarction and pulmonary embolism.

The use of intraoperative opioids can result in an exaggerated response to pain (hyperalgesia) and contribute to an exacerbation of pain after surgical procedures.Opioids are commonly given intraoperative, not in response to pain, but in response to hyperdynamic cardiovascular states. Esmolol is a short acting beta 1 antagonist that can be used to treat/prevent hyperdynamic states during surgery. More importantly, esmolol has been shown to have central antihyperalgesic effects that might contribute to a reduction in postoperative pain. It is therefore conceivable that the use of intraoperative esmolol instead of opioids to avoid hyperdynamic states during surgery can result in lower postoperative pain. Since postoperative pain can substantially affect postoperative quality of recovery, it is also conceivable that the use of intraoperative esmolol might result in an improved postoperative quality of recovery to surgical patients.

The main objective of the current study is to examine the effect of intraoperative esmolol on postoperative quality of recovery. A secondary objective is to examine the effect of esmolol on postoperative pain.

Significance: Postoperative pain after ambulatory surgery has been shown to be poorly managed in The United States. The goal of this study is to investigate if a change in the intraoperative pharmacologic management of patients undergoing ambulatory surgery can improve their postoperative quality of recovery and pain.

The research question is; does the use of intraoperative esmolol improve postoperative quality of recovery after ambulatory surgery? Does the use of intraoperative esmolol improve postoperative pain after ambulatory surgery?

The hypotheses of this study is; does the use of intraoperative esmolol improves postoperative quality of recovery after ambulatory surgery. The use of intraoperative esmolol reduces postoperative pain after ambulatory surgery.

DETAILED DESCRIPTION:
We propose a randomized double blinded placebo controlled clinical trial. Healthy females undergoing outpatient surgery will be recruited . Before surgery patients will be tested for pain sensitivity and threshold using a Pathway Pain & sensory evaluation system (Medoc, Dunham, NC).Subjects will randomized using a computer generated table of random numbers to two groups: Active (Esmolol 0.5 mg/kg followed by an infusion of 5-15 mcg/kg/min titrated to keep heart rate between 50 and 70 BPM) or control (same volume of normal saline).The infusion will be discontinued at the end of the surgical procedure. Subjects will receive a standard anesthetic regimen: Induction (2 mg versed, 1-2mg /kg propofol and 0.6mg/kg of rocuronium), maintenance (Sevoflurane titrated to a Bispectral index between 40-60 and fentanyl 50 mcg q 10 minutes to maintain blood pressure within 20% of baseline value. Patients will receive at the end of surgery ondansetron 4 mg IV to prevent nausea and/or vomiting. The postoperative analgesic regimen will also be standardized with hydromorphone 0.4 mg every 15 minutes to treat pain greater than 4/10 (scale where 0 means no pain and 10 means the worst possible pain) and hydrocodone 10 mg/acetaminophen 325 for pain control after discharge. Patients will receive ephedrine 5 mg q5minutes if blood pressure is lower than 40% baseline or if the heart rate is less than 40 beats per minute. Before hospital discharge patients will again be tested for pain sensitivity and threshold using a Pathway Pain & sensory evaluation system (Medoc, Dunham, NC).

The primary outcome will be a validated instrument to measure postoperative quality of recovery (QoR-40) that will be administered to patients by an investigator unaware of group allocation at 24 hours after the surgery.Other outcomes to be evaluated include; postoperative pain sensitivity and threshold, postoperative opioid consumption, postoperative pain, time to meet discharge criteria using a validated instrument (PADDS).

ELIGIBILITY:
Inclusion Criteria:

- Female patients Undergoing outpatient hysteroscopic myomectomy surgery ASA PS I and II Age between 18 and 64 years Fluent in English

Exclusion Criteria:

History of allergy to beta-blocker History of chronic opioid use Pregnant patients BMI greater than 35 History of EKG abnormalities or cardiac arrhythmias Beta-blocker medication usage.

Dropout criteria: Patient or surgeon request, Conversion of the surgery from laparoscopic to open.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Womens Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Esmolol | .9 Normal Saline
Started | 35 | 35
Completed | 29 | 29
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esmolol | .9 Normal Saline | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 38 [31 to 45] | 41 [32 to 50] | 39 [31 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
BMI (kg/m^2) [Median (Full Range); unit: (kg/m^2)] — BMI is the abbreviation for body mass index which is represented by the following:
  (kg/m^2)
  (kg/m^2) | 23 [22 to 29] | 24 [23 to 26] | 24 [22 to 29]
Intraoperative Fentanyl (mcg) [Median (Full Range); unit: micrograms] | 100 [50 to 150] | 100 [50 to 150] | 100 [50 to 150]
Surgical Duration [Median (Full Range); unit: Minutes] | 82 [67 to 99] | 72 [66 to 83] | 77 [67 to 99]
American Society of Anesthesiologist Classification [Number; unit: participants] — The grading system is to evaluate the degree of a patient's physical state before undergoing anesthetic procedure. 1-6 1 being healthy patient and 6 being brain dead.
  participants
    ASA Class 1 | 12 | 11 | 23
    ASA Class 2 | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Qor-40 at 24 Hours Postoperative
Description: Quality of recovery questionnaire score at 24 hours after surgery. Quality of recovery score 24 hours after the surgical procedure.Score of 40 is poor recovery and a score of 200 is good recovery.
  Time frame for this evaluation is 24 hours after the surgical procedure
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale 40 low-200 high
Arm/Group | Esmolol | .9 Normal Saline
Number analyzed (Participants) | 29 | 29
units on a scale 40 low-200 high | 179 [171 to 190] | 182 [173 to 189]
Statistical Analysis 1: Comparison: Esmolol vs .9 Normal Saline; Test type: Superiority or Other; p = .82, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Postoperative Opioid Consumption
Description: The total amount of opioid consumed by subject at 24 hours after surgery measured in IV morphine equivalents.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: IV mg of morpine equivalents
Arm/Group | Esmolol | .9 Normal Saline
Number analyzed (Participants) | 29 | 29
IV mg of morpine equivalents | 2.5 [0 to 6] | 0 [0 to 4]
Statistical Analysis 1: Comparison: Esmolol vs .9 Normal Saline; Test type: Superiority or Other; p = .05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Post Operative Pain Reported by the Subject.
Description: Post operative pain reported by the subject as determined as area under the numeric rating scale for pain versus time curve in the post anesthesia care unit ( score*min).Numeric rating scale for pain on a scale of 0-10 (0 is no pain and 10 is high pain) versus time curve in the post anesthesia care unit ( score * min). A higher value indicates more pain over 24 hours.The range is 0 pain to x time in minutes x hour ( 60-1440 minutes) . The pain scores were collected at 15 minute intervals from the time of admission to the PACU to 24 hours after the surgical procedure. The area under the NRS pain scale versus time curve was calculated using the trapezoidal method as an indicator of pain burden during early recovery (Graph Pad Prism ver 5.03, Graph Pad Software INC.
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: (pain score * minutes ) in the PAC U
Arm/Group | Esmolol | .9 Normal Saline
Number analyzed (Participants) | 29 | 29
(pain score * minutes ) in the PAC U | 218 [90 to 270] | 150 [45 to 240]
Statistical Analysis 1: Comparison: Esmolol vs .9 Normal Saline; Test type: Superiority or Other; p = .14, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Esmolol | .9 Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 10/29 | 10/29
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmolol (N=29) | .9 Normal Saline (N=29)
Nausea (Gastrointestinal disorders) | 9 (9) | 10 (10)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No